CLINICAL TRIAL: NCT03709095
Title: Sprint Interval Training During Rehabilitation After Spinal Cord Injury
Acronym: SprintSCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SprintSCI
Record Dates: First submitted 2018-10-11; First posted 2018-10-17 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Spinal Cord Injuries; Rehabilitation; Exercise
Keywords: Inpatient Rehabilitation; Sprint interval training; Exercise; Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Participants were randomized to one of two groups: (A) sprint interval training (SIT) or (B) moderate intensity continuous training (MICT).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate Intensity Continuous Training (Active Comparator): Training was performed three times a week for five weeks. Each session began with a 2 minute warm up, and concluded with a 3 minute cool down. Following the warm-up, participants performed 20 minutes of arm cycling at a self-selected cadence at 45-65% of their peak power output. Total training duration was 25 mins.
  Interventions: Other: moderate intensity continuous training
- Sprint Interval Training (Experimental): The SIT protocol was adopted from Gillen and colleagues (See Ref), and consisted of 3 x 20 second "all-out" efforts at ≥ 100% of an individuals peak power output. Each sprint was interspersed by 120 seconds of active recovery at 10% of an individuals peak power output. Total training duration was 10 mins.
  Interventions: Other: Sprint interval training

INTERVENTIONS:
Other: Sprint interval training — Participants utilized the arm ergometer for improving aerobic exercise capacity
  Arms: Sprint Interval Training
Other: moderate intensity continuous training — Participants utilized the arm ergometer for improving aerobic exercise capacity
  Arms: Moderate Intensity Continuous Training

SUMMARY:
Immediately following a spinal cord injury (SCI), patients are admitted to inpatient rehabilitation where they undergo physical reconditioning in preparation for a return to home setting. The current standard of practice for aerobic training is performing arm-ergometry for 25 mins at a frequency of three times per week. Given the move towards shortened length of stay during inpatient rehabilitation, performing MICT can consume a considerable amount of therapy time. Sprint interval training (SIT) has been shown to elicit similar improvements in physical capacity, despite a reduced time commitment to MICT. However, there are no controlled trials comparing the effects of SIT to MICT in individuals with SCI undergoing inpatient rehabilitation. The primary aim of this study was to investigate the efficacy of a five-week, thrice weekly 10 min SIT program and compare outcome measures to a traditional 25 minute MICT program on the arm-ergometer in individuals with SCI undergoing inpatient clinical rehabilitation. It was hypothesized that five weeks of SIT and MICT would induce similar changes in maximal and sub-maximal exercise performance, self-efficacy for exercise, and exercise enjoyment, despite large differences in training volume and time commitment. It was also hypothesized that SIT would be well tolerated and elicit higher levels of cardiovascular strain than MICT.

ELIGIBILITY:
Inclusion Criteria:

* Participants with sub-acute spinal cord injury (time since injury: 14 - 182 days)
* Undergoing inpatient rehabilitation
* Aged 18-65 years
* Injury level at the second cervical vertebrae (C2) or below

Exclusion Criteria:

- Unable to perform arm-ergometry training

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Change in peak power output | Change in peak power output from baseline to 5 weeks
  maximum amount of power produced during a graded exercise test on the arm-ergometer
Change in sub-maximal arm-ergometry | Change in sub-maximal arm-ergometry from baseline to 5 weeks
  Participants performed three 5-minute steady state workloads on the arm-ergometer at power outputs corresponding to RPE's of 8, 10 and 12. Participants were given a minimum of 2 minutes, and a maximum of 5 minutes of rest in between each workload.

SECONDARY OUTCOMES:
Cardiovascular Responses | Throughout each week of training (Week 1,Week 2, Week 3, Week4, Week 5)
  Monitored heart rate throughout each training session
Perceptual Responses | Throughout each week of training (Week 1,Week 2, Week 3, Week4, Week 5)
  Monitored ratings of perceived exertion throughout each training session
Change in self-efficacy for exercise | Change in self-efficacy from baseline to 5 weeks
  Using a self-reported questionnaire, participants rated how confident they are with regards to performing and carrying out regular physical activities and exercises.
Exercise Satisfaction | Measured only at the end of the intervention (5 weeks)
  Participants completed the Physical Activity Enjoyment Scale (PACES) in order to asses the level of enjoyment with the training intervention they received.
Pain perceptions | Measured only at the end of the intervention (5 weeks)
  Through a questionnaire, participants rated how much shoulder pain, bodily pain, and physical discomfort they typically experience throughout the day and how much pain they experienced with the intervention they were allocated to.

CONTACTS AND LOCATIONS:
Overall Officials: Audrey L Hicks, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gillen JB, Martin BJ, MacInnis MJ, Skelly LE, Tarnopolsky MA, Gibala MJ. Twelve Weeks of Sprint Interval Training Improves Indices of Cardiometabolic Health Similar to Traditional Endurance Training despite a Five-Fold Lower Exercise Volume and Time Commitment. PLoS One. 2016 Apr 26;11(4):e0154075. doi: 10.1371/journal.pone.0154075. eCollection 2016. PMID 27115137
- [Background] Hicks AL, Martin KA, Ditor DS, Latimer AE, Craven C, Bugaresti J, McCartney N. Long-term exercise training in persons with spinal cord injury: effects on strength, arm ergometry performance and psychological well-being. Spinal Cord. 2003 Jan;41(1):34-43. doi: 10.1038/sj.sc.3101389. PMID 12494319
- [Background] Nightingale TE, Metcalfe RS, Vollaard NB, Bilzon JL. Exercise Guidelines to Promote Cardiometabolic Health in Spinal Cord Injured Humans: Time to Raise the Intensity? Arch Phys Med Rehabil. 2017 Aug;98(8):1693-1704. doi: 10.1016/j.apmr.2016.12.008. Epub 2017 Jan 13. PMID 28089898
- [Background] Astorino TA, Thum JS. Within-session responses to high-intensity interval training in spinal cord injury. Disabil Rehabil. 2018 Feb;40(4):444-449. doi: 10.1080/09638288.2016.1260648. Epub 2016 Dec 8. PMID 27930890